CLINICAL TRIAL: NCT06833853
Title: CTC-EXPRESS: A Prospective Observational Study for CTC Expression and cfDNA/RNA Assessment in Metastatic Breast Cancer
Brief Title: A Study for CTC Expression and cfDNA/RNA Assessment in Metastatic Breast Cancer Patients
Acronym: CTC-EXPRESS
Status: Not yet recruiting | Type: Observational
Sponsor: Menarini Silicon Biosystems, INC (Industry)
Responsible Party: Sponsor
Other Study IDs: CTC-EXPRESS
Record Dates: First submitted 2025-02-10; First posted 2025-02-19 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Metastatic Breast Cancer (MBC)
Keywords: CTC; cfDNA; cfRNA
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- HR+/HER2- subjects before starting 1st line therapy: Subjects will receive CTC enumeration, CTC HER2, ER, PD-L1 expression and, and MSearch cfDNA/RNA assessments at baseline and first restaging as part of standard of care. Subjects will have additional cfDNA/RNA tests at week 4, and 8.
- Triple negative starting any line of therapy, HR+/HER2-, and HER2+ starting ≥2nd line therapy: Subjects will receive CTC enumeration, and CTC HER2, ER, PD-L1 expression minimally before each restaging visit, and cfDNA/RNA assessments at baseline and first restaging as part of standard of care.

SUMMARY:
The purpose of this research is to learn if the CellSearch Circulating Tumor Cells (CTC) test can help doctors in making decisions about treatment and monitoring of breast cancer. The test consists of diagnostic CTC counts (enumeration) and expression of biomarkers Human Epidermal growth factor Receptor 2 (HER2), Estrogen Receptor (ER), and programmed death-ligand 1 (PD-L1) and cell free DNA/RNA (cfDNA/RNA) analysis.

DETAILED DESCRIPTION:
A prospective, multicenter, observational study of CellSearch CTC enumeration, CTC HER2, ER, and PD-L1 expression, and MSearch cfDNA/RNA results in subjects with histologically proven MBC. Treatment for MBC will be chosen and performed by treating physicians/providers. Eligible subjects will be enrolled after signing the ICF. Subjects will receive CTC enumeration, CTC HER2, ER, PD-L1 expression and, and MSearch cfDNA/RNA assessments at baseline and first restaging as part of Standard of Care (SoC). Subjects will receive any additional cfDNA/RNA assessments as part of research collection. For all subjects 4 to 6 tubes will be collected at baseline and minimally before the first restaging visit. For any subsequent restaging visits a total of 3 to 4 tubes will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Invasive breast cancer with radiographic and/or clinical evidence of advanced metastatic or unresectable disease.
* HR+/HER2 negative or triple negative (TN) subjects prior to starting first line therapy or beyond in the metastatic setting.

OR HER2+ subjects prior to starting second line therapy or beyond in the metastatic setting.

* Subject must have the CTC HER2, ER, PD-L1, and cfDNA/RNA tests ordered during routine patient care.
* Age > 18 years.

Exclusion Criteria:

* Participant is pregnant.
* Inability to provide blood samples based on the judgment of the treating physician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Advanced/metastatic breast cancer of following subtypes/lines of systemic therapy in metastatic setting:
  * Estrogen Receptor (ER)+/Human Epidermal growth factor Receptor 2 (HER2) - or Triple Negative (TN) patients prior to starting any line of systemic therapy
  * HER2+ patients prior to starting 2nd line or later therapy
Sampling Method: Probability Sample
Enrollment: 187 (Estimated)
Dates: Start 2025-10-15 (Estimated); Primary Completion 2027-10-01 (Estimated); Study Completion 2029-03-01 (Estimated)

PRIMARY OUTCOMES:
The percentage of subjects for which the providers indicated positive impact of the cfDNA/RNA, CTC enumeration, and CTC expression results. | 3-4 months
  The percentage of subjects for which the providers indicated positive impact on treatment decisions or response assessment of the cfDNA/RNA, CTC enumeration, and CTC expression assessments.CTC enumeration, CTC biomarker expression, and cfDNA/RNA results in subjects with MBC.

SECONDARY OUTCOMES:
The correlation of CTC expression and tissue immunohistochemistry (IHC)/In Situ Hybridization (ISH) results for HER2, ER, and PD-L1. | 1 month
The correlation of CTC expression and cfDNA/RNA results for HER2, ER, and PD-L1. | 3-4 months
The correlation of CTC HER2, ER and PD-L1 expression with response to therapy and progression free survival (PFS). | 24 months
The correlation of cfDNA/RNA genomic alterations with response to therapy and PFS. | 24 months
The correlation of early cfDNA/RNA dynamics with response to therapy and PFS in 1st line Hormone Receptor (HR) +/HER2- MBC. | 24 months
The correlation of CTC enumeration results with PFS. | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Marija Balic, MD, PhD, MBA, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Magee Womens Hospital, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided